CLINICAL TRIAL: NCT07156851
Title: Observational BELgian Registry of Implanted EV-ICD to Evaluate Parameters and Complications of the New Device in Real World Settings
Acronym: BELIEVE
Status: Not yet recruiting | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Jean-Benoît Le Polain de Waroux, Coordinating Principal Investigator, AZ Sint-Jan AV
Other Study IDs: BELIEVE
Record Dates: First submitted 2025-03-18; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Implantable Cardioverter Defibrillator (ICD)
Keywords: Extravascular implantable cardioverter-defibrillator; EV-ICD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to follow all patients implanted with extravascular implantable cardioverter-defibrillators (EV-ICDs) in Belgium throughout the lifetime of the devices. The main goal of the study is to keep track of:

* all parameters of the device
* complications
* arrhythmia detection and therapy delivery
* clinical endpoints (quality of life, cardiac and infectious events) Participants who underwent or will undergo an EV-ICD implantation as part of their regular medical care will be asked if data can be collected from their medical record. No additional tasks are required for the study.

DETAILED DESCRIPTION:
The BELIEVE registry (BELgian registry of Implanted EV-ICDs to Evaluate parameters and complications) is a multicenter, observational registry designed to gather real-world data on the use of extravascular implantable cardioverter-defibrillators (EV-ICDs) in Belgium. This new generation of ICD technology offers the potential advantages of both subcutaneous (S-ICD) and transvenous (TV-ICD) devices, with the lead placed under the sternum. This position enables pacing capabilities and more accurate arrhythmia detection while aiming to minimize lead-related complications seen in previous ICD systems.

Given the relatively recent introduction of EV-ICDs, it is essential to monitor their performance and clinical outcomes in routine clinical settings. While initial trials have demonstrated feasibility and safety, real-world data are crucial for understanding long-term efficacy, complication rates, therapy effectiveness, device longevity, and overall patient outcomes. The BELIEVE registry was therefore established to support this need, offering a structured framework to follow patients over time and improve clinical practice related to EV-ICDs.

The registry is both retrospective and prospective, non-randomized, and will include all patients in Belgium who undergo (or have undergone) an EV-ICD implantation-regardless of whether the procedure was successful. Participating centers will aim to enroll an initial cohort of 100 patients over a 4-year period, although the number of patients and study duration may be extended. The total planned study period is 15 years, with patients followed throughout the life of their device.

Inclusion criteria are broad: participants must be at least 18 years old, have had or be scheduled for an EV-ICD implantation (even if unsuccessful), and must provide informed consent. Patients who did not undergo any part of the implantation procedure are excluded.

Data will be collected at baseline, during the procedure, and during scheduled follow-up visits (at 1-3 months, 6 months, and then at least annually). Information will include demographic and clinical characteristics, medical history, device data, arrhythmia detection, therapy delivery, programming changes, complications, and patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Previous or planned EV-ICD implantation (successful or not)
* Informed consent signed

Exclusion Criteria:

* Patients who did not undergo any step of the implantation procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent or will undergo an EV-ICD implantation in Belgium, whether successful or not, can be included in this registry.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2040-07-01 (Estimated); Study Completion 2040-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of delivered therapies (ATP and shocks) | Lifetime of the device (up to 15 years)
  Total number of therapies delivered by the device, including antitachycardia pacing and shocks (Unit: count)
Proportion of delivered therapies that were appropriate | Lifetime of the device (up to 15 years)
  Percentage of therapies delivered by the device that were adjudicated as appropriate (i.e., delivered for true ventricular arrhythmia).
Proportion of delivered therapies that were successful | Lifetime of the device (up to 15 years)
  Percentage of therapies delivered by the device that successfully terminated the targeted ventricular arrhythmia.
Tracking procedural and device-related complications | Lifetime of the device (up to 15 years)
  Tracking procedural and device-related complications during the lifetime of the device

SECONDARY OUTCOMES:
Change in sensing amplitude over time | Lifetime of the device (up to 15 years)
  Change in device-recorded sensing amplitude (in mV) from implantation to follow-up visits.
Change in pacing threshold over time | Lifetime of the device (up to 15 years)
  Change in pacing threshold (in Volt) measured during device follow-up from implantation to 15 years.
Change in lead impedance over time | Lifetime of the device (up to 15 years)
  Change in lead impedance (in Ohm) from implantation to 15 years of follow-up.
Change in battery longevity estimates over time | Lifetime of the device (up to 15 years)
  Change in estimated battery longevity (in years) as reported by the device at each follow-up visit.
Accuracy of arrhythmia detection by the device | Lifetime of the device (up to 15 years)
  Proportion of arrhythmia episodes correctly classified by the device (%)
Summary of device reprogramming | Lifetime of the device (up to 15 years)
  Summary of every device reprogramming including reason for changes
Number of participants with major adverse cardiac events (MACE) | Lifetime of the device (up to 15 years)
  Number of participants experiencing major adverse cardiac events, including cardiovascular death, hospitalization for heart failure, myocardial infarction, or stroke.
Number of participants with device-related infections | Lifetime of the device (up to 15 years)
  Number of participants with infections requiring antibiotic treatment or device/system extraction.
Number of participants reporting device-related complaints | Lifetime of the device (up to 15 years)
  Number of participants reporting device-related symptoms or complaints (e.g., inappropriate shocks, pain at device site).